CLINICAL TRIAL: NCT00600782
Title: Immunogenicity and Safety of GSK Biologicals' Candidate Tuberculosis (TB) Vaccine (692342) When Administered to Healthy Adults Aged 21 to 40 Years.
Brief Title: Immunogenicity and Safety of a Candidate Tuberculosis (TB) Vaccine Given to Healthy Adults in a TB-endemic Region
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 110347
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Tuberculosis (TB); Tuberculosis Vaccines
Keywords: Tuberculosis vaccine
MeSH Terms: conditions — Tuberculosis | interventions — Vaccines

ARMS (1):
- Group A (Experimental): These subjects were further stratified into 3 groups according to the size of their PPD skin test reactions
  Interventions: Biological: GSK Biologicals' Candidate Tuberculosis (TB) Vaccine (692342)

INTERVENTIONS:
Biological: GSK Biologicals' Candidate Tuberculosis (TB) Vaccine (692342) — Intramuscular injection, 2 doses at 0, 1 month

SUMMARY:
This study will assess the safety and immunogenicity of a GSK Biologicals' candidate TB vaccine administered at 0, 1 months to healthy adults living in a TB-endemic region. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the Investigator believes that they can and will comply with the requirements of the protocol.
* A male or female between, and including, 21 and 40 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to any study procedure.
* Free of obvious health problems as established by medical history and clinical examination before enrolment into the study.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.
* No evidence of pulmonary pathology as confirmed by chest X-ray.
* Clinically normal laboratory values for creatinine, ALT, AST and complete blood count.
* Seronegative for human immunodeficiency virus-1 (HIV-1).
* No history of extrapulmonary TB.
* Subjects must have the appropriate PPD skin reactivity (induration measured at 48 to 72 hours after PPD skin test administration).

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* History of previous administration of experimental Mycobacterium tuberculosis vaccines.
* History of previous exposure to experimental products containing MPL or QS21.
* Administration of any immunoglobulins, any immunotherapy and/or any blood products within the three months preceding the first dose of study vaccination, or planned administrations during the study period.
* Participation in another experimental protocol during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency. Subjects who describe a first-degree relative with clearly documented autoimmune disease will be excluded
* History of any acute or chronic illness or medication that, in the opinion of the Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
* Any chronic drug therapy to be continued during the study period, with the exception of vitamins and/or dietary supplements, birth control pills, anti-histamines for seasonal allergies, SSRIs.
* History of any neurologic disorders or seizures.
* History of allergic reactions or anaphylaxis to previous immunisations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of chronic alcohol consumption and/or drug abuse which in the investigators opinion would put the subject at risk.
* Major congenital defects.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2008-02-05 (Actual); Primary Completion 2008-12-19 (Actual); Study Completion 2008-12-19 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of solicited local and general symptoms | During the 7-day follow-up period following vaccination after each vaccine dose
Occurrence, intensity and relationship to vaccination of unsolicited symptoms | During the 30-day follow-up period following vaccination after each vaccine dose
Occurrence and relationship to vaccination of serious adverse events | During the entire study period
Haematological and biochemical levels | At protocol defined time points

SECONDARY OUTCOMES:
Analysis of cytokine expression by M72-specific CD4+/CD8+ T cells by means of invitro flow cytometry | At protocol defined time points
Antibody titres to M72 measured by ELISA | At protocol defined time points

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Worcester, Western Province, South Africa

REFERENCES:
- [Background] Day CL, Tameris M, Mansoor N, van Rooyen M, de Kock M, Geldenhuys H, Erasmus M, Makhethe L, Hughes EJ, Gelderbloem S, Bollaerts A, Bourguignon P, Cohen J, Demoitié MA, Mettens P, Moris P, Sadoff JC, Hawkridge A, Hussey GD, Mahomed H, Ofori-Anyinam O, Hanekom WA. Induction and regulation of T-cell immunity by the novel tuberculosis vaccine M72/AS01 in South African adults. PMID:23306546